CLINICAL TRIAL: NCT02843308
Title: Building Community-Academic Partnerships for the Evidence-Based Treatment of Hoarding Disorder
Brief Title: Enhancing Treatment of Hoarding Disorder With Personalized In-Home Sorting and Decluttering Practice
Acronym: BITS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Carolyn Rodriguez, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36788; K23MH092434 (NIH)
Record Dates: First submitted 2016-07-20; First posted 2016-07-25 (Estimated); Results first posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Hoarding Disorder; Hoarding; Clutter
Keywords: hoarding disorder; hoarding; clutter
MeSH Terms: conditions — Hoarding Disorder; Hoarding; Speech Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate Treatment (Experimental): Facilitated group therapy with behavioral practice; 18 weeks
  Interventions: Behavioral: Facilitated group therapy with behavioral practice; 18 weeks
- Delayed Treatment (Experimental): Facilitated group therapy with behavioral practice; 18 weeks (after a 18-20 week delay)
  Interventions: Behavioral: Facilitated group therapy with behavioral practice; 18 weeks

INTERVENTIONS:
Behavioral: Facilitated group therapy with behavioral practice; 18 weeks — Facilitated group therapy for hoarding disorder with behavioral practice

SUMMARY:
The proposed study aims to investigate the efficacy of adding in-home decluttering practice to Buried in Treasures Workshop (BIT) facilitated group treatment for hoarding disorder.

DETAILED DESCRIPTION:
Patients participate in Buried in Treasures Workshop (BIT) that has been shown to improve symptoms of hoarding disorder. The investigators hypothesize that adding in-home decluttering practice to the BIT workshop will decrease hoarding symptoms and level of clutter over time.

ELIGIBILITY:
Inclusion Criteria for Individuals with Hoarding Disorder:

1. Age 18 to 70 years
2. Either gender and all ethno-racial groups
3. Physically healthy male or non-pregnant female.
4. Hoarding Disorder primary condition
5. Willing and able to understand and complete consent and study procedures
6. English speaking

Exclusion Criteria for Individuals with Hoarding Disorder:

1. Current or past history of bipolar, psychotic or eating disorders, substance dependence, or substance abuse in the last year.
2. Clinically at risk of suicide with Columbia Suicide Severity Rating Scale (C-SSRS) Suicidal Ideation Subscale of 4 or higher (i.e. suicidal intent without specific plan)
3. Major medical or neurological conditions that increase the risk of participation or that would prevent completing assigned behavioral practice tasks.
4. Unable or unwilling to allow study staff into home for home assessment
5. Currently at high risk for eviction
6. Animal hoarding or squalor

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2020-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Rodriguez, M.D., Ph.D., Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wheaton MG, Varias AD, Sandhu T, Munoz Rodriguez PA, Mukunda P, Filippou-Frye M, Millen A, Lombardi A, van Roessel P, Raila H, Anderson K, Linkovski O, Mahnke A, Sanchez C, McCarthy E, Wright B, Mibenge C, Rico Y, Righi S, Halsey C, Torio L, Asgari S, Qiu T, Garcia G, Jo B, Belofsky B, Shuer LJ, Frost RO, Rodriguez CI. Randomized waitlist-controlled trial of buried in treasures facilitated support groups and in-home uncluttering (BIT+) for hoarding disorder. J Psychiatr Res. 2024 Aug;176:58-67. doi: 10.1016/j.jpsychires.2024.05.055. Epub 2024 May 30. PMID 38843580
- See also: Rodriguez Lab Website — http://med.stanford.edu/rodriguezlab.html
- See also: Dr. Carolyn Rodriguez Faculty Page — https://med.stanford.edu/profiles/carolyn-rodriguez?tab=bio

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Immediate Treatment | Delayed Treatment
Started | 21 | 20
Completed | 18 | 19
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Treatment | Delayed Treatment | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.29 (12.06) | 58.45 (8.41) | 56.37 (10.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 27
  Male | 6 | 8 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 12
  Not Hispanic or Latino | 15 | 14 | 29
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Met and Exceeded Response Criteria of the Saving Inventory-Revised (SI-R)
Description: The SI-R is a 23-item questionnaire with 3 sub-scales for difficulty discarding, excessive clutter, and compulsive acquisition.
  The total score ranges from 0 to 92. The greater the score, the more severe the hoarding symptoms. Total score higher than 41 shows significant difficulty with clutter.
  For the acquisition subscale, items 2 (reverse score), 9, 11, 14, 16, 18 and 21 are summed together. The subscale ranges from 0 to 28 and score greater than 13 indicates difficulty with excessive acquisition.
  For the difficulty discarding subscale, items 4(reverse score), 6, 7, 13, 17, 19, 23 are summed together. The subscale ranges from 0 to 28 and score greater than 13 indicates difficulty with discarding.
  For the clutter subscale, items 1, 3, 5, 8, 10, 12, 15, 20, 22 are summed together. The subscale ranges from 0 to 36 and score greater than 15 indicates difficulty with accumulated clutter.
  Response was defined as at least a 14 point change (pre-post) in the total score.
Time Frame: Change from baseline (pre-treatment) to week 18 (post-treatment) the Immediate Treatment Arm/Group and change from baseline (pre-treatment at 18 weeks) to 36 weeks (post-treatment) for the Delayed Treatment Arm/Group
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Treatment | Delayed Treatment
Number analyzed (Participants) | 18 | 19
Participants | 9 | 13

ADVERSE EVENTS:
Time Frame: Baseline (pre-treatment) up to 18 weeks for the Immediate Treatment Arm/Group and up to 36 weeks for the Delayed Treatment Arm/Group
Arm/Group | Immediate Treatment | Delayed Treatment
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 0/21 | 0/20

LIMITATIONS AND CAVEATS:
Several limitations deserve consideration (see paper Wheaton et al., 2024). Although this is the first trial of BIT+ to include a control group, the group was limited to waiting list (which controlled for the passage of time) and did not include another credible treatment comparator. As a result, other potential confounding variables such as placebo effects and attention from the research team were not controlled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-11-11): https://cdn.clinicaltrials.gov/large-docs/08/NCT02843308/Prot_SAP_000.pdf
  • Informed Consent Form (2020-05-31): https://cdn.clinicaltrials.gov/large-docs/08/NCT02843308/ICF_001.pdf